CLINICAL TRIAL: NCT07289906
Title: Measurement of Mass Change in Serum Albumin Compared to Serum Lactic Acid as Predictive Tool for Sepsis Prognosis in Non Surgical ICU Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: MD241/2025
Record Dates: First submitted 2025-12-05; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Prognosis Prediction of Sepsis in Icu Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Diagnostic Test: Mass change in serum albumin — study aims to assess the accuracy of measurement of mass change in serum albumin compared to serum lactic acid as predictive tool for sepsis prognosis in nonsurgical ICU patients
  Other Names: Serum lactate

SUMMARY:
This study aims to assess the reliability of measurement of mass change in serum albumin compared to serum lactic acid as predictive tool for sepsis prognosis in nonsurgical ICU patients

DETAILED DESCRIPTION:
This study explores the prognostic value of mass change in serum albumin compared to serum lactic acid levels in non-surgical ICU patients with sepsis. While serum lactate is an established marker of tissue hypo-perfusion and a predictor of sepsis outcomes, serum albumin is less frequently used for dynamic monitoring, although it is known to correlate with severity and mortality

Measurements:

Data Collection:

A-Baseline Data on ICU Admission:

1. Demographics: age, sex
2. Comorbidities (e.g., diabetes, hypertension, chronic kidney disease)
3. Initial hemodynamic parameters (BP-HR-SO2-ECG-UOP-TEMP-RR)
4. diagnosis of sepsis involves recognising signs of infection plus organ dysfunction according to SSC and sepsis -3

   A- Search about source of infection by:
   * History of present illness about main complain.
   * clinical examination
   * investigation a. labs (CBC (containing TLC and platlets), CRP, Procal, BloodGases (containing serum lactate), Urea, serum Creatinine, TotaL bilirubin, Urine Analysis, Pan culture, AST, ALT) b-imaging (chest x.ray) B- organ dysfunction Defined as increase increase in SOFA (Sequential Organ Failure Assessment) score >=2 points from baseline.

   SOFA Score range:

   0-6: low risk of organ failure 7-12: moderate risk >12: high risk of mortality
5. initial reading of serum albumin in admission (T0)
6. initial reading of albumin creat ratio (ACR)as tool for measuring albumin in urine Patients with severe albuminuria will be excluded from the study

Daily measurements:

1. Average of 24 HR (BP, HR, SO2, TEMP, RR,)
2. CBC, CRP, serum urea, serum creatinine, Total bilirubin, serum Albumin, blood gases (containing serum lactate)

3-24HR Fluid balance.

* ACR will be measured every 3days during study to predict any abnormal increase in albumin loss in urine

C- Daily recordings:

1. SOFA score.
2. mass changes in serum albumin (T0-T1, T1-T2, T3-T2……...ETC).
3. serum lactate.
4. vasopressor use.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 year 70 years. Diagnosis of sepsis according to survival sepsis campaign(SSC). Patients admitted for medical (non-surgical) conditions.

Exclusion Criteria:

* Chronic liver disease or cirrhosis. Hyperalbuminuria (ex: nephrotic syndrome, nephritic syndrome). Terminal illness with an expected survival of less than 24 hours. Refusal or inability to obtain informed consent from patients or their care givers.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A prospective cohort study is planned, aiming to enroll a minimum of 40 patients. The sample size calculation is based on findings from Mahashabde et al. (2024), which reported that the predictive accuracy of serum lactase for septic shock at admission had an AUC ROC of 0.96, while serum albumin had an AUC ROC of 0.323. The anticipated incidence of septic shock is 42%, as reported in the EPIC ill study (2019). The sample size was calculated to achieve 100% statistical power with a significance level (alpha) of 0.05.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-09-28 (Actual); Primary Completion 2026-09-28 (Estimated); Study Completion 2026-09-28 (Estimated)

PRIMARY OUTCOMES:
Comparative value between mass change in serum albumin and serum lactate in prediction of sepsis prognosis (discharge or mortality) | 12 months
  Knowing Which is more accurate in predicting the prognosis of sepsis between mass change in serum albumin and serum lactic acid in non surgical icu patients

SECONDARY OUTCOMES:
Duration of vasopressor use and its correlation to prognosis of sepsis. | 12months
  If long duration of using vasopressor correlate with prognosis of sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Alaa E Mohamed Hassen, Prof, Study Director — Department of anesthesia ,Intensive Care and pain management
Locations (1):
- Hospitals ofAin shams university, Cairo, Elabasya, Egypt

IPD SHARING:
Plan to Share IPD: No